CLINICAL TRIAL: NCT04614974
Title: Initiation of Acid Suppression Therapy Prospective Outcomes for Laryngomalacia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow recruitment due to few eligible patients
Sponsor: Reema Padia (Other)
Responsible Party: Sponsor-Investigator, Reema Padia, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20090193
Record Dates: First submitted 2020-10-22; First posted 2020-11-04 (Actual); Results first posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Laryngomalacia; Gastro Esophageal Reflux
Keywords: Laryngomalacia; Symptom improvement; Famotidine; Speech Language Therapy
MeSH Terms: conditions — Laryngomalacia; Gastroesophageal Reflux; Communication Disorders | interventions — Famotidine; Speech Therapy

STUDY DESIGN:
Intervention Model Description: Experimental, open-label randomized control trial
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Speech Language Therapy Alone (Experimental): Patients in this group will receive a routine swallowing evaluation by a speech language pathologist. Patient caregivers will fill out the Infant Gastroesophageal Reflux Questionnaire (I-GERQ-R) and the Pittsburgh Airway Symptom Score (PASS) the day of the appointment and at the 3-month follow up appointment.
  Interventions: Other: Speech Language Therapy
- Speech Language Therapy and Acid Suppression Therapy (Active Comparator): Patients in this group will receive a routine swallowing evaluation by a speech language pathologist and famotidine (acid suppression therapy). Patient caregivers will fill out the Infant Gastroesophageal Reflux Questionnaire (I-GERQ-R) and the Pittsburgh Airway Symptom Score (PASS) the day of the appointment and at the 3-month follow up appointment.
  Interventions: Drug: Famotidine; Other: Speech Language Therapy

INTERVENTIONS:
Drug: Famotidine — Famotidine will be prescribed based on patients' weight. Caregivers will purchase this medication and dosage will be given to families in easy-to-understand language.
  Arms: Speech Language Therapy and Acid Suppression Therapy
Other: Speech Language Therapy — Speech Language Therapy (feeding therapy) will be provided by a speech language pathologist to assess feeding and swallowing.

SUMMARY:
Laryngomalacia (LM) is the most common cause of stridor in infants. Symptoms of gastroesophageal reflux (GER) are often seen in the setting of LM; therefore, acid suppression therapy (AST) has been empirically used in the management of this disorder. The investigators recently performed a retrospective chart review assessing improvement of airway and dysphagia symptoms, weight gain, and need for surgery with AST. It was found that there was a similar improvement between LM severity groups and most patients received AST (96.6%). It is unclear if these improvements are due to AST or natural resolution of the disease. With heightened concerns of side effects related to AST in infants, particularly among those born prematurely, judicious use of these medications is needed. The investigators are now performing a prospective study looking at the outcome differences in patients with laryngomalacia who are evaluated by speech language therapy (SLP) alone versus those with SLP evaluation and acid suppression therapy (famotidine).

DETAILED DESCRIPTION:
Purpose: To determine the outcome differences in patients 6 months and younger with laryngomalacia and dysphagia who are evaluated by speech language therapy (SLP) alone versus those with both SLP evaluation and acid suppression therapy (AST) (famotidine)

Hypothesis: There will be no differences in outcomes between those that had SLP alone versus those that had both SLP and AST.

Laryngomalacia (LM) is the most common cause of stridor in infants. Symptoms of gastroesophageal reflux (GER) are often seen in the setting of LM; therefore, acid suppression therapy (AST) has been empirically used in the management of this disorder. However, there is no gold standard in treating mild and moderate LM patients and therefore this study will help establish guidelines for treatment.

A medical chart review will be performed to assess airway and dysphagia symptom improvement from consult to the 3-month follow up appointment and then up to a year. The Pittsburgh Airway Symptom Score (PASS) questionnaire and the Infant Gastroesophageal Reflux Questionnaire (I-GERQ-R) will be given to families at the consult and at the 3-month follow up appointment for caregiver assessment. The physician will then perform the standard procedures at the clinic appointment. The Flexible Laryngoscopy Findings sheet will be filled out in conjunction with the clinic procedures for objective data. The surveys will then be scored to determine true GERD (score >=16) and severe laryngomalacia (LM) (RED questions on the PASS), which would further exclude these patients. There are 12 total questions on the I-GERQ-R. On the PASS, questions 1 & 2 are in the GREEN category and signifies mild LM, YELLOW signifies moderate LM, and RED is severe LM. On the PASS questionnaire, "Yes" to either #1 or #2 and nothing else is mild LM, "yes" to at least one #3-5 and none of #6-10 is moderate LM, and "yes" to any of the #6-10" indicates severe LM. There are 10 total questions on the PASS. Mild and moderate LM patients will be block randomized the day before the appointment to receive speech language therapy alone or speech language therapy with famotidine (Pepcid). Both treatments are standard of care in these patients. Speech language therapy (feeding therapy) is part of the normal clinic visit for LM patients. These patients will then be re-evaluated at their follow up appointment in 3 months (+/- 1 month). The families will take the PASS and I-GERQ-R surveys again to determine LM severity.

Initially, primary outcome #2 was "Dysphagia symptom score change from consult (baseline) to 3 month follow-up appointment." This is the same as the original secondary outcome measure #6 "Infant Gastroesophageal Reflux Questionnaire (I-GERQ-R) score change from consult (baseline) to 3 month follow-up appointment" (I-GERQ-R is the dysphagia symptom score used in this study). Therefore, these were consolidated to a single primary outcome measure "Infant Gastroesophageal Reflux Questionnaire (I-GERQ-R) score change from consult (baseline) to 3 month follow-up appointment." This change was made after study and data collection completion, at the time of results reporting.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients ages 0 to 6 months who do need meet the criteria at the initial appointment for supraglottoplasty
* Seen in University of Pittsburgh Medical Center (UPMC) Children's Hospital of Pittsburgh (CHP) Otolaryngology Department
* Laryngomalacia without prolonged (>20 seconds) cyanosis, apnea, nor failure to thrive.

Exclusion Criteria:

* Children over the age of 6 months old will be excluded from participation.
* Premature infants (<37 weeks gestation)
* Patients with lung disease.
* Laryngomalacia with prolonged (>20 seconds) cyanosis, apnea, and failure to thrive
* Sleep induced laryngomalacia
* Patients with craniofacial abnormalities
* Patients with a syndrome
* Patients with additional airway abnormalities, seen before or at consult
* Patients with symptoms that necessitate surgery
* Patients with a prior cardiac surgery
* Patients with AST prescribed prior to the initial otolaryngology consult.

Ages: 0 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reema Padia, MD, Principal Investigator — Division of Pediatric Otolaryngology, Children's Hospital of Pittsburgh
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosbe KW, Kenna MA, Auerbach AD. Extraesophageal reflux in pediatric patients with upper respiratory symptoms. Arch Otolaryngol Head Neck Surg. 2003 Nov;129(11):1213-20. doi: 10.1001/archotol.129.11.1213. PMID 14623753
- [Background] Hartl TT, Chadha NK. A systematic review of laryngomalacia and acid reflux. Otolaryngol Head Neck Surg. 2012 Oct;147(4):619-26. doi: 10.1177/0194599812452833. Epub 2012 Jun 27. PMID 22745201
- [Background] Bibi H, Khvolis E, Shoseyov D, Ohaly M, Ben Dor D, London D, Ater D. The prevalence of gastroesophageal reflux in children with tracheomalacia and laryngomalacia. Chest. 2001 Feb;119(2):409-13. doi: 10.1378/chest.119.2.409. PMID 11171716
- [Background] Landry AM, Thompson DM. Laryngomalacia: disease presentation, spectrum, and management. Int J Pediatr. 2012;2012:753526. doi: 10.1155/2012/753526. Epub 2012 Feb 27. PMID 22518182
- [Background] Thompson DM. Laryngomalacia: factors that influence disease severity and outcomes of management. Curr Opin Otolaryngol Head Neck Surg. 2010 Dec;18(6):564-70. doi: 10.1097/MOO.0b013e3283405e48. PMID 20962644
- [Derived] Shaffer AD, Balogun Z, Tobey ABJ, Maguire RC, Simons JP, Dohar JE, Mccoy JL, Rushchak MV, Padia R. Acid Suppression in Mild-Moderate Laryngomalacia Without GERD: A Randomized Controlled Trial. Laryngoscope. 2026 Jan;136(1):471-478. doi: 10.1002/lary.32471. Epub 2025 Aug 5. PMID 40762274

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only infant patients were considered enrolled.
Period: Overall Study
Arm/Group | Speech Language Therapy Alone | Speech Language Therapy and Acid Suppression Therapy
Started | 34 | 31
Completed | 20 | 20
Not Completed | 14 | 11
Not completed — Lost to Follow-up | 14 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Speech Language Therapy Alone | Speech Language Therapy and Acid Suppression Therapy | Total
Number analyzed (Participants) | 34 | 31 | 65
Age, Continuous [Median (Full Range); unit: Months] — Age at initial consult
  Months | 2.3 [0.5 to 6.8] | 2.3 [0.2 to 6.2] | 2.3 [0.2 to 6.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 23 | 17 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 28 | 24 | 52
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 31 | 29 | 60
  Unknown or Not Reported | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Airway Symptom Score Change From Consult (Baseline) to 3 Month Follow-up Appointment
Description: Score change from pre to post surveys on the Pittsburgh Airway Symptom Score (PASS) questionnaire. The PASS is on a scale from 0-10 with a higher score indicating a worse outcome. This outcome will be assessed at the consult and the 3 month follow-up appointment.
Time Frame: 3 months
Population: Follow-up PASS was completed by 20/34 (59%) in the speech language therapy alone group and 20/31 (65%) of the speech language therapy and acid suppression therapy group.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Speech Language Therapy Alone | Speech Language Therapy and Acid Suppression Therapy
Number analyzed (Participants) | 20 | 20
score on a scale
  Baseline | 3 [2 to 5] | 3 [1 to 5]
  Change from baseline to 3 months | -2 [-5 to 2] | -1 [-4 to 1]
Statistical Analysis 1: Comparison: Speech Language Therapy Alone vs Speech Language Therapy and Acid Suppression Therapy; Test type: Superiority; p = 0.3, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Infant Gastroesophageal Reflux Questionnaire (I-GERQ-R) Score Change From Consult (Baseline) to 3 Month Follow-up Appointment
Description: Score change from pre to post survey on the I-GERQ-R. There are 12 questions on the surveys on a scale of 0-42. A higher score indicates a worse outcome. Those with a score of >=16 on this survey at the initial consult are excluded from the study, indicating true gastroesophageal reflux disease (GERD). This outcome will be assessed at the consult and the 3 month follow-up appointment.
Time Frame: 3 months
Population: Follow-up I-GERQ-R was completed by 20/34 (59%) in the speech language therapy alone group and 20/31 (65%) of the speech language therapy and acid suppression therapy group. However, 1 participant in the speech language therapy alone group only completed questions 1-6 of the I-GERQ-R and therefore was not included in analysis of total I-GERQ-R scores.
Measure: Median (Full Range); unit: score on scale
Arm/Group | Speech Language Therapy Alone | Speech Language Therapy and Acid Suppression Therapy
Number analyzed (Participants) | 19 | 20
score on scale
  Baseline | 12 [6 to 15] | 10 [5 to 15]
  Change from baseline to 3 months | -4 [-12 to 11] | -3 [-11 to 9]
Statistical Analysis 1: Comparison: Speech Language Therapy Alone; Test type: Superiority; p = 0.8, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Change in Prevalence of Airway Symptoms From Consult up to 1 Year Assessed Via Electronic Medical Chart Review
Description: Change in prevalence of airway symptoms from consult up to 1 year assessed via electronic medical chart review. Notes from the Department of Otolaryngology will be reviewed which include reported symptoms from caregivers and symptoms seen upon exam. Airway symptoms included periods of apnea, chest wall retractions, cyanosis, stridor, noisy breathing, and increased respiratory rate.
Time Frame: 1 year
Population: 15 participants in the speech language therapy alone group and 21 participants in the speech language therapy and acid suppression therapy group had a follow-up otolaryngology clinic visit within 1 year of initial consult.
Measure: Count of Participants; unit: Participants
Arm/Group | Speech Language Therapy Alone | Speech Language Therapy and Acid Suppression Therapy
Number analyzed (Participants) | 15 | 21
Participants
  Apnea: Symptom absent at consult and follow-up | 14 | 20
  Apnea: Symptom present at consult, absent at follow-up | 0 | 0
  Apnea: Symptom absent at consult, present at follow-up | 0 | 1
  Apnea: Symptom present at consult and follow-up | 1 | 0
  Chest Wall Retractions: Symptom absent at consult and follow-up | 12 | 19
  Chest Wall Retractions: Symptom present at consult, absent at follow-up | 2 | 1
  Chest Wall Retractions: Symptom absent at consult, present at follow-up | 0 | 1
  Chest Wall Retractions: Symptom present at consult and follow-up | 1 | 0
  Cyanosis: Symptom absent at consult and follow-up | 15 | 21
  Cyanosis: Symptom present at consult, absent at follow-up | 0 | 0
  Cyanosis: Symptom absent at consult, present at follow-up | 0 | 0
  Cyanosis: Symptom present at consult and follow-up | 0 | 0
  Stridor: Symptom absent at consult and follow-up | 1 | 4
  Stridor: Symptom present at consult, absent at follow-up | 5 | 7
  Stridor: Symptom absent at consult, present at follow-up | 1 | 0
  Stridor: Symptom present at consult and follow-up | 8 | 10
  Noisy Breathing: Symptom absent at consult and follow-up | 2 | 1
  Noisy Breathing: Symptom present at consult, absent at follow-up | 2 | 10
  Noisy Breathing: Symptom absent at consult, present at follow-up | 0 | 1
  Noisy Breathing: Symptom present at consult and follow-up | 11 | 9
  Increased respiratory rate: Symptom absent at consult and follow-up | 15 | 21
  Increased respiratory rate: Symptom present at consult, absent at follow-up | 0 | 0
  Increased respiratory rate: Symptom absent at consult, present at follow-up | 0 | 0
  Increased respiratory rate: Symptom present at consult and follow-up | 0 | 0
Statistical Analysis 1: Comparison: Speech Language Therapy Alone; Noisy breathing pre/post; Test type: Other; p = 0.5, McNemar
Statistical Analysis 2: Comparison: Speech Language Therapy and Acid Suppression Therapy; Noisy breathing pre/post; Test type: Other; p = 0.01, McNemar
Statistical Analysis 3: Comparison: Speech Language Therapy Alone; Stridor pre/post; Test type: Other; p = 0.2, McNemar
Statistical Analysis 4: Comparison: Speech Language Therapy and Acid Suppression Therapy; Stridor pre/post; Test type: Superiority; p = 0.02, McNemar
Statistical Analysis 5: Comparison: Speech Language Therapy Alone; Chest wall retractions pre/post; Test type: Other; p = 0.5, McNemar
Statistical Analysis 6: Comparison: Speech Language Therapy and Acid Suppression Therapy; Chest wall retractions pre/post; Test type: Other; p = 1.0, McNemar
Statistical Analysis 7: Comparison: Speech Language Therapy Alone; Apnea pre/post; Test type: Other; p = 1.0, McNemar

4. Primary Outcome: Change in Prevalence of Dysphagia Symptoms From Consult up to 1 Year Assessed Via Electronic Medical Chart
Description: Change in prevalence of dysphagia symptoms from consult up to 1 year assessed via electronic medical chart review. Notes from the Department of Otolaryngology will be reviewed which include reported symptoms from caregivers and symptoms seen upon exam. Dysphagia symptoms included choking, coughing, gagging with feeds and/or emesis after feeds.
Time Frame: 1 year
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Speech Language Therapy Alone | Speech Language Therapy and Acid Suppression Therapy
Number analyzed (Participants) | 15 | 21
Participants
  Emesis: Symptom absent at consult and follow-up | 3 | 7
  Emesis: Symptom present at consult, absent at follow-up | 5 | 7
  Emesis: Symptom absent at consult, present at follow-up | 2 | 1
  Emesis: Symptom present at consult and follow-up | 5 | 6
  Choking: Symptom absent at consult and follow-up | 9 | 11
  Choking: Symptom present at consult, absent at follow-up | 5 | 3
  Choking: Symptom absent at consult, present at follow-up | 0 | 3
  Choking: Symptom present at consult and follow-up | 1 | 4
  Coughing: Symptom absent at consult and follow-up | 7 | 9
  Coughing: Symptom present at consult, absent at follow-up | 7 | 5
  Coughing: Symptom absent at consult, present at follow-up | 0 | 5
  Coughing: Symptom present at consult and follow-up | 1 | 2
  Gagging: Symptom absent at consult and follow-up | 13 | 17
  Gagging: Symptom present at consult, absent at follow-up | 2 | 2
  Gagging: Symptom absent at consult, present at follow-up | 0 | 2
  Gagging: Symptom present at consult and follow-up | 0 | 0
Statistical Analysis 1: Comparison: Speech Language Therapy Alone; Emesis pre/post; Test type: Other; p = 0.5, McNemar
Statistical Analysis 2: Comparison: Speech Language Therapy and Acid Suppression Therapy; Emesis pre/post; Test type: Other; p = 0.07, McNemar
Statistical Analysis 3: Comparison: Speech Language Therapy Alone; Choking pre/post; Test type: Superiority; p = 0.06, McNemar
Statistical Analysis 4: Comparison: Speech Language Therapy and Acid Suppression Therapy; Choking pre/post; Test type: Other; p = 1.0, McNemar
Statistical Analysis 5: Comparison: Speech Language Therapy Alone; Coughing pre/post; Test type: Other; p = 0.02, McNemar
Statistical Analysis 6: Comparison: Speech Language Therapy and Acid Suppression Therapy; Coughing pre/post; Test type: Other; p = 1.0, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Speech Language Therapy and Acid Suppression Therapy; Gagging pre/post; Test type: Other; p = 1.0, McNemar

5. Secondary Outcome: Weight (kg/Month) From Consult up to 1 Year
Description: Weight change in kilograms per month assessed from medical chart review from consult up to 1 year
Time Frame: 1 year
Population: 20 patients in the speech language therapy alone group and 27 patients in the speech therapy and acid suppression therapy group had weights available in the electronic medical record from at least 1 follow-up appointment with any specialty within 1 year.
Measure: Median (Full Range); unit: kg/month
Arm/Group | Speech Language Therapy Alone | Speech Language Therapy and Acid Suppression Therapy
Number analyzed (Participants) | 20 | 27
kg/month | 0.62 [0.27 to 1.04] | 0.56 [0.24 to 0.84]
Statistical Analysis 1: Comparison: Speech Language Therapy Alone vs Speech Language Therapy and Acid Suppression Therapy; Test type: Superiority; p = 0.3, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Number of Participants With the Need for Supraglottoplasty Surgery (Escalation of Treatment) up to 1 Year
Description: The need for escalation of treatment with supraglottoplasty surgery will be assessed through medical chart review up to 1 year.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Speech Language Therapy Alone | Speech Language Therapy and Acid Suppression Therapy
Number analyzed (Participants) | 34 | 31
Participants | 2 | 1
Statistical Analysis 1: Comparison: Speech Language Therapy Alone vs Speech Language Therapy and Acid Suppression Therapy; Test type: Superiority; p = 1.0, Fisher Exact

7. Secondary Outcome: Number of Participants With the Need for Acid Suppression Therapy Medication (Famotidine) From Speech Language Therapy Alone Group From the Day After the Consult up to 1 Year
Description: The speech language therapy alone group will be assessed for the need for a prescription for acid suppression therapy (famotidine) from the day after the consult up to 1 year.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Speech Language Therapy Alone
Number analyzed (Participants) | 34
Participants | 6

8. Secondary Outcome: Number of Participants With Each Type of Laryngomalacia (Types 1-3) Found on the Flexible Laryngoscopy Procedure at the Consult
Description: All patients will be scoped with a flexible laryngoscopy at the initial consult and the type of laryngomalacia (Types 1-3) will be noted. Participants are reported for each type of laryngomalacia noted at the initial consent. Participants can have more than one type of laryngomalacia. Type 1 is characterized by anterior/medial collapse of supra-arytenoid mucosa. Type 2 is characterized by short aryepiglottic folds. Type 3 is characterized by posterior collapse of epiglottis. None are considered better/worse outcomes.
Time Frame: At initial consult
Measure: Count of Participants; unit: Participants
Arm/Group | Speech Language Therapy Alone | Speech Language Therapy and Acid Suppression Therapy
Number analyzed (Participants) | 34 | 31
Participants
  Type 1-Anterior/medial collapse of supra-arytenoid mucosa | 29 | 27
  Type 2-Short AE folds | 24 | 19
  Type 3- Posterior collapse of epiglottis | 4 | 4

9. Secondary Outcome: Number of Participants With the Need for a Different Acid Suppression Therapy Medication (Other Than Famotidine) From the Day After the Consult up to the 3 Month Follow up Appointment
Description: Both groups will be assessed for the need for a different acid suppression therapy medication (other than famotidine) from the day after the consult up to the 3 month follow up appointment.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Speech Language Therapy Alone | Speech Language Therapy and Acid Suppression Therapy
Number analyzed (Participants) | 34 | 31
Participants | 0 | 2

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Speech Language Therapy Alone | Speech Language Therapy and Acid Suppression Therapy
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/31
Serious Adverse Events (participants affected / at risk) | 3/34 | 3/31
Other Adverse Events (participants affected / at risk) | 7/34 | 8/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Speech Language Therapy Alone (N=34) | Speech Language Therapy and Acid Suppression Therapy (N=31)
Hospital admission for viral infection (Infections and infestations) | 2 (4) | 1 (1)
Pediatric intensive care unit admission for respiratory distress following supraglottoplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Inguinal hernia with incarceration requiring surgery (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Hospital admission for seizure (Nervous system disorders) | 0 (0) | 2 (2)
Hospital admission for monitoring post-motor vehicle accident (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Speech Language Therapy Alone (N=34) | Speech Language Therapy and Acid Suppression Therapy (N=31)
Emergency department visit broken femur (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Emergency department visit eczema and skin yeast infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Emergency department visit viral syndrome (Infections and infestations) | 5 (6) | 5 (7)
Emergency department visit constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Emergency department post-fall (General disorders) | 0 (0) | 2 (2)
Emergency department visit abscess (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Emergency department visit tachypnea, fussiness, spitting up (Gastrointestinal disorders) | 0 (0) | 1 (1)
Emergency department visit seizures (Nervous system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-14): https://cdn.clinicaltrials.gov/large-docs/74/NCT04614974/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-12): https://cdn.clinicaltrials.gov/large-docs/74/NCT04614974/ICF_001.pdf